CLINICAL TRIAL: NCT04030936
Title: Knowledge Regarding Diagnosis of Molar Incisor Hypomineralization Among Dental Interns in Faculty of Dentistry Cairo University
Brief Title: Knowledge Regarding Diagnosis of MIH Among Dental Interns in Faculty of Dentistry Cairo University
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Norhan Yahia Mohamed Mahmoud, Dentist, Ministry of health, Egypt, Cairo University
Other Study IDs: umnaz
Record Dates: First submitted 2019-07-21; First posted 2019-07-24 (Actual); Last update posted 2019-09-13 (Actual); Status verified 2019-09

CONDITIONS: Molar Incisor Hypomineralization
Keywords: MIH, knowledge , Molar Incisor Hypomineralization
MeSH Terms: conditions — Molar Hypomineralization

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
assessment of knowledge of dental interns regarding diagnosis of MIH among Group of interns in faculty of dentistry Cairo university

DETAILED DESCRIPTION:
The study will be done in faculty of dentistry Cairo university in form of survey with data being gathered via a questionnaire. The survey was conducted among the dental interns

ELIGIBILITY:
Inclusion Criteria:

* any nationality both gender

Exclusion Criteria:

* interns who refuse to participate

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: dental interns in faculty of dentistry Cairo university
Sampling Method: Probability Sample
Enrollment: 190 (Estimated)
Dates: Start 2019-09 (Estimated); Primary Completion 2020-07 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
knowledge regarding diagnosis of MIH | one year
  questionnaire (yes or no and Multiple choice questions)

IPD SHARING:
Plan to Share IPD: Undecided